CLINICAL TRIAL: NCT04756778
Title: Relationship Between Indexed Aortic Area and Aortic Diameter in Bicuspid Aortic Valve Aortopathy: A Retrospective Cohort Study
Brief Title: Indexed Aortic Area in Bicuspid Aortic Valve Aortopathy
Status: Completed | Type: Observational
Sponsor: St. George's Hospital, London (Other)
Responsible Party: Principal Investigator, Metesh Acharya, Mr Metesh Acharya, St. George's Hospital, London
Other Study IDs: IAAinBAVAneurysms2021
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Thoracic Aortic Aneurysm; Bicuspid Cardiac Valve
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Aortic surgery +/- aortic valve replacement — Replacement of aneurysmal proximal thoracic aorta +/- replacement of diseased bicuspid aortic valve

SUMMARY:
This study aims to determine the relationship between the cross-sectional aortic area/patient height ratio (indexed aortic area) and absolute aortic diameter in proximal thoracic aortic aneurysms associated with a bicuspid valve. This will shed light on whether aneurysms with smaller diameters than those recommended for surgical intervention by guidelines are still at risk of aortic complications attending an abnormally high indexed aortic area.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* First-time surgery
* Bicuspid aortic valve confirmed
* Thoracic aortic aneurysm involving aortic root or ascending aorta

Exclusion Criteria:

* No available pre-operative cross-sectional imaging
* Re-do surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients undergoing first-time surgery for a BAV-related aneurysm involving the aortic root and/or ascending aorta, between 2010-2016 at our institution
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Median aortic diameters in aneurysms | Data collection period from 27th January 2017 - 15th May 2017
  As above
Cross-sectional aortic area/patient height ratio in aneurysms | Data collection period from 27th January 2017 - 15th May 2017
  Calculation of indexed aortic area in aneurysms
Proportion of aneurysms with cross-sectional aortic area/patient height ratio >10 cm2/m | Data collection period from 27th January 2017 - 15th May 2017
  Proportion of aneurysms with an abnormal indexed aortic area
Median cross-sectional aortic area/patient height ratio for aneurysms with diameter <4.0 cm, 4.0-4.5 cm, 4.5-5.0 cm, 5.0-5.5 cm and >5.5 cm | Data collection period from 27th January 2017 - 15th May 2017
Median aortic diameter corresponding to aneurysms with IAA >10 cm2/m | Data collection period from 27th January 2017 - 15th May 2017

CONTACTS AND LOCATIONS:
Locations (1):
- St. George's Hospital, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No